CLINICAL TRIAL: NCT04436874
Title: Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Dai Ethnic Group as Donor Source in Terms of Treatment Efficacy and Pathogenic Mechanisms
Brief Title: Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease
Acronym: FMT-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yinglei Miao, Clinical professor，Director of Gastroenterology, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMT-IBD-190923
Record Dates: First submitted 2020-06-02; First posted 2020-06-18 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Fecal Microbiota Transplantation
Keywords: Ulcerative Colitis; Crohn's disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Han ethnic-UC (Experimental): Ulcerative colitis subjects will be treated with bacterial solution from Han ethnic by endoscopy
  Interventions: Device: endoscopy
- Han ethnic-CD (Experimental): Crohn's disease subjects will be treated with bacterial solution from Han ethnic by endoscopy
  Interventions: Device: endoscopy
- Dai ethnic-UC (Experimental): Ulcerative colitis subjects will be treated with bacterial solution from Dai ethnic by endoscopy
  Interventions: Device: endoscopy
- Dai ethnic-CD (Experimental): Crohn's disease subjects will be treated with bacterial solution from Dai ethnic by endoscopy
  Interventions: Device: endoscopy

INTERVENTIONS:
Device: endoscopy — transplant infusion of feces from healthy donors into affected subjects

SUMMARY:
Fecal microbiota transplantation (FMT), defined as infusion of feces from healthy donors to affected subjects, is a method to restore a balanced gut microbiota and has attracted great interest in recent years due to its efficacy and ease of use.

DETAILED DESCRIPTION:
FMT is now recommended as the most effective therapy for CDI not responding to standard therapies1.Recent studies have suggested that dysbiosis is associated with a variety of disorders, and that FMT could be a useful treatment. Randomized controlled trial has been conducted in a number of disorders including ulcerative colitis (UC). Our study is aims to Fecal microbiota transplantation in the treatment of Inflammatory Bowel Disease, the role of selection of the Dai ethnic group as donor source in terms of treatment efficacy and pathogenic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years inclusive (no limit on gender)
* Confirmed diagnosis of ulcerative colitis for > 3 months, according to established clinical,endoscopic and histologic criteria
* Currently active mild-moderate ulcerative colitis, as measured by a Mayo score of 4-10, in which endoscopy sub-score ≥ 1 and physician's global assessment sub-score ≤ 2
* Written informed consent obtained.

Exclusion Criteria:

* Subjects who are unable to give consent or who have conditions rendering them incapable to answer questionnaires or provide samples.
* Females who are pregnant or actively trying to fall pregnant
* Subjects unwilling to practice an effective method of contraception throughout the study period
* Subjects defined as in remission by the investigator
* Evidence or history of toxic megacolon
* Isolated proctitis < 5 cm
* A diagnosis of Crohn's Disease or indeterminate colitis
* Subjects with perianal disease (e.g. fistulae, pre-existing fissures)
* Significant gastrointestinal surgery e.g. colon resection, colectomy :Minor gastrointestinal surgery will be reviewed on a case by case basis by the investigator;Regarding appendicectomy, only exclude patients who had appendicectomy < 3 months ago)
* Subjects taking antimicrobials (antibiotics, antifungals, antivirals) for any reason, including antibiotics for ulcerative colitis, in the preceding 4 weeks
* Subjects who are steroid dependent and requiring > 20mg prednisone or > 9mg budesonide daily at the time of enrolment
* Subjects who have recently taken or are actively taking or expected to require prohibited medication/s during the study period including follow-up. These include:Rectal therapy including corticosteroid, 5-aminosalicylate within 2 weeks before first FMT;Treatment with biologic agents e.g. infliximab, adalimumab, vedolizumab, within 12 weeks before first FMT;Treatment with other major immunosuppressant agents including calcineurin inhibitors, anti-neoplastic agents, lymphocyte depleting biological agents within 12 weeks before first FMT;Probiotic therapy within 4 weeks before first FMT;Experimental / trial drug protocol involvement within 12 weeks before first FMT;Anti-mycobacterial (TB or MAC) therapy within 4 weeks before first FMT

Allowed concomitant medications:

The following drugs are allowed as long as the dose is stable preceding first FMT for the noted time:

* oral 5-aminosalicylates (stable dose for 4 weeks)
* thiopurines and methotrexate (on medication for ≥ 90 days and dose stable for 4 weeks)
* oral prednisolone (dose ≤ 20mg daily and stable for 2 weeks) During the study, subjects should remained on the same dose of oral 5-aminosalicylate, thiopurine, and methotrexate. For oral prednisolone, dose must be tapered at a rate up to 2.5mg per week so that subjects would be steroid-free by week 8.

Prohibited medications:

The following drugs for are prohibited for the noted time:

* Rectal therapies including corticosteroid, 5-aminosalicylate (for 2 weeks before first FMT and during study period)
* Antibiotics, antibiotics, antifungals, antivirals, probiotic or prebiotic preparations (for 4 weeks before first FMT and during study period)
* Rectal therapies including corticosteroid, 5-aminosalicylate (for 2 weeks before first FMT and during study period)
* Biological therapies or calcineurin inhibitors (for 12 weeks before first FMT and during study period)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
steroid-free clinical remission and endoscopic remission | 3 years
  The primary outcome is a composite of steroid-free clinical remission together with endoscopic remission or response at week 6, defined as defined as a total Mayo score of ≤2 points with no individual sub-score >1 point, and at least a 1 point reduction from baseline in the endoscopy sub-score

SECONDARY OUTCOMES:
Steroid-free clinical remission | 3 years
  defined as combined Mayo sub-scores of 1 or less for rectal bleeding plus stool frequency
Steroid-free clinical response | 3 years
  defined as either a decrease of 3 points or more on the Mayo score, a 50% or greater reduction from baseline in combined rectal bleeding plus stool frequency Mayo sub-scores, or both
Steroid-free endoscopic response | 3 years
  defined as a Mayo endoscopy sub-score of 1 or less, with a reduction of at least 1 point from baseline
microbiological change | 3 years
  Changes in microbial composition (including bacteriome, virome and fungome), function and metabolite
Change in microbiome of stool | 3 years
  Change in microbiome of stool (including bacteriome, virome and fungome)
Difference in microbiome compared between subjects in different treatment arm | 3 years
  Difference in microbiome (including bacteriome, virome and fungome) compared between subjects in different treatment arm
Proportion of microbiome | 3 years
  Proportion of microbiome (including bacteriome, virome and fungome) derived from recipient, donor or both in subjects who received FMT
Difference in microbiome compared between subjects who have weight loss and those do not have weight loss | 3 years
  Difference in microbiome (including bacteriome, virome and fungome) compared between subjects who have weight loss and those do not have weight loss
Microbial factors that are associated with percentage of body weight loss | 3 years
  Microbial factors (including bacteriome, virome and fungome) that are associated with percentage of body weight loss
Trans-kingdom correlation of microbial engraftment after FMT between bacteriome, virome and fungome | 3 years
  Trans-kingdom correlation of microbial engraftment after FMT between bacteriome, virome and fungome

CONTACTS AND LOCATIONS:
Overall Officials: Y L Miao, doctor, Study Director — First Affiliated Hospital of Kunming Medical University
Locations (1):
- Endoscopy, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No